CLINICAL TRIAL: NCT02773030
Title: A Phase 1b/2a Multicenter, Open-label, Dose-escalation Study to Determine the Maximum Tolerated Dose, Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of CC-220 as Monotherapy and in Combination With Other Treatments in Subjects With Multiple Myeloma
Brief Title: A Study to Determine Dose, Safety, Tolerability, Drug Levels, and Efficacy of CC-220 Monotherapy, and in Combination With Other Treatments in Participants With Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-MM-001; U1111-1182-9200 (Registry Identifier: WHO); 2016-000860-40 (EudraCT Number)
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; Pharmacokinetics; Safety; Efficacy; CC-220; Relapsed and refractory multiple myeloma; Dexamethasone; Daratumumab; Bortezomib; Newly diagnosed multiple myeloma; Newly diagnosed multiple myeloma transplant non-eligible
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — iberdomide; Dexamethasone; Calcium Dobesilate; daratumumab; Bortezomib; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort A: CC-220 Monotherapy - Part 1 (Experimental): Oral CC-220 at dose specified by cohort dose level from Day 1-21 of each 28-day cycle
  Interventions: Drug: CC-220
- Cohort B: CC-220 in combination with Dexamethasone (DEX) - Part 1 (Experimental): Oral CC-220 at dose specified by cohort dose level from Day 1-21 of each 28-day cycle.
  For subjects ≤ 75 years old, oral DEX 40 mg on Days 1, 8, 15, and 22 of each 28-day cycle. For subjects >75 years old, DEX will be administered at 20 mg on Days 1, 8,15, and 22 of each 28-day cycle. Subjects who surpass the age of 75 years while on treatment may be switched to the 20 mg QD dosage based on the investigator's best judgment.
  Interventions: Drug: CC-220; Drug: Dexamethasone
- Cohort D: CC-220 in combination with Dexamethasone - Part 2 (Experimental): Oral CC-220 at Recommended Phase 2 dose (RP2D) from Day 1-21 of each 28-day cycle
  For subjects ≤ 75 years old, oral DEX 40 mg on Days 1, 8, 15, and 22 of each 28-day cycle. For subjects >75 years old, DEX will be administered at 20 mg on Days 1, 8, 15, and 22 of each 28-day cycle
  Interventions: Drug: CC-220; Drug: Dexamethasone
- Cohort E: CC-220 with DEX and daratumumab (DARA) - Part 1 (Experimental): Oral CC-220 at dose specified by cohort dose level from Day 1-21 of each 28-day cycle.
  Oral DEX for subjects ≤ 75 years old at 40 mg on Days 1, 8, 15, and 22 of each 28-day cycle. For subjects >75 years old, oral DEX at 20 mg on Days 1, 8, 15, and 22 of each 28-day cycle.
  Intravenous DARA at dose 16mg/kg on Days 1, 8, 15, and 22 at cycle 1-2, Days 1, 15 at cycle 3-6, and Day 1 at cycle ≥7 of each 28-day cycle.
  Once the MTD and/or RP2D is determined in Cohort E (CC-220Dd), subjects will be enrolled at a dose of Subcutaneous DARA at 1800 mg over 3 to 5minutes on Days 1, 8, 15,and 22 at cycle 1-2 of a 28-day cycle, Days1, and 15 at cycle 3-6 of a 28-day cycle, and Day1 at cycle ≥7 of each 28-day cycle.
  Interventions: Drug: CC-220; Drug: Dexamethasone; Drug: Daratumumab
- Cohort F: CC-220 with DEX and bortezomib - Part 1 (Experimental): Oral CC-220 at dose specified by cohort dose level from Day 1-14 of each 21-day cycle.
  Oral DEX for subjects ≤ 75 years old at 40 mg on Days 1, 8, and 15 of each 21-day cycle. For subjects >75 years old, oral DEX at 20 mg on Days 1, 8, and 15 of each 21-day cycle.
  Subcutaneous BTZ at dose 1.3 mg/m^2 on Days 1, 4, 8 and 11 at cycle 1-8, and Days 1, and 8 at cycle ≥9 of each 21-day cycle.
  Interventions: Drug: CC-220; Drug: Dexamethasone; Drug: Bortezomib
- Cohort G1: CC-220 in combination with CFZ and DEX - Part 1 (Experimental): Oral CC-220 at dose specified by cohort dose level from Day 1-21 of each 28-day cycle
  Intravenous (IV) CFZ (Carfilzomib)administered at a starting dose of 20 mg/m2 on C1D1; and at a dose specified by cohort dose level thereafter on days 1, 8, and 15 of each 28-day cycle.
  Oral DEX (Dexamethasone) on Days 1, 8, 15, and 22 of each 28-day cycle. For subjects ≤ 75 years old, the DEX dose will be 40 mg. For subjects > 75 years old, the DEX dose will be 20 mg
  Interventions: Drug: CC-220; Drug: Dexamethasone; Drug: Carfilzomib
- Cohort G2 - CC-220 in combination with CFZ and DEX - Part 1 (Experimental): Oral CC-220 at dose specified by cohort dose level from Day 1-21 of each 28-day cycle.
  Intravenous (IV) CFZ administered at a starting dose of 20 mg/m2 on C1D1 and C1D2; and at a dose level specified by cohort dose level thereafter Days 1, 2, 8, 9, 15, 16 of each 28-day cycle.
  Oral DEX on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle. The DEX dose will be 20 mg.
  Interventions: Drug: CC-220; Drug: Dexamethasone; Drug: Carfilzomib
- Cohort I: CC-220 in combination with DEX in post BCMA RRMM - Part 2 (Experimental): Oral CC-220 at Recommended Phase 2 dose (RP2D) from Day 1-21 of each 28-day cycle
  Oral DEX 40 mg on Days 1, 8, 15, and 22 of each 28-day cycle. For subjects >75 years old, oral DEX will be administered at 20 mg on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: CC-220; Drug: Dexamethasone
- Cohort J1: CC-220 in combination with DEX and BTZ in NDMM - Part 2 (Experimental): Oral CC-220 at 1.0mg, 1.3mg or 1.6mg administered at cycles 1 to 8 on Days 1 to 14 of each 21-day cycle and cycles ≥ 9 on Days 1 to 21 of each 28-day cycle.
  Oral DEX at Cycles 1 to 8, 20 mg (≤ 75 years old) or 10 mg (> 75 years old) on Days 1, 2, 4, 5, 8, 9, 11 and 12 of each 21-day cycle and Cycles ≥ 9, 40 mg (≤ 75 years old) or 20 mg (> 75 years old) on Days 1, 8, 15, and 22 of each 28-day cycle.
  Subcutaneous BTZ at dose 1.3 mg/m2 on Days 1, 4, 8 and 11 at Cycle 1-8 of each 21-day cycle.
  Interventions: Drug: CC-220; Drug: Dexamethasone; Drug: Bortezomib
- Cohort J2: CC-220 in combination with DEX and BTZ in NDMM - Part 2 (Experimental): Oral CC-220 at Recommended Phase 2 Dose from Day 1-14 of each 21-day cycle.
  Oral DEX at 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) for Cycles 1 to 6 on Days 1, 2, 4, 5, 8, 9, 11 and 12 of a 21-day cycle.
  Subcutaneous BTZ at dose 1.3 mg/m2 on Days 1, 4, 8 and 11 at Cycle 1-6 of each 21-day cycle.
  Interventions: Drug: CC-220; Drug: Dexamethasone; Drug: Bortezomib
- Cohort K: CC-220 with DEX and DARA in NDMM and not autologous stem cell transplant eligible - Part 2 (Experimental): Oral CC-220 at 1.0mg, 1.3mg or 1.6mg from Days 1-21 of each 28-day cycle.
  Oral DEX 40 mg on Days 1, 8, 15, and 22 of each 28-day cycle. For subjects >75 years old, oral DEX will be administered at 20 mg on Days 1, 8, 15, and 22 of each 28-day cycle.
  Subcutaneous DARA at 1800 mg over 3 to 5minutes on Days 1, 8, 15, and 22 at cycle 1-2 of a 28-day cycle, Days1, and 15 at cycle 3-6 of a 28-day cycle, and Day1 at cycle ≥7 of each 28-day cycle.
  Interventions: Drug: CC-220; Drug: Dexamethasone; Drug: Daratumumab
- Cohort C: CC-220 Monotherapy in RRMM - Part 2 (Experimental): CC-220 at dose specified by cohort dose level from Day 1-21 of each 28-day cycle.
  Interventions: Drug: CC-220

INTERVENTIONS:
Drug: CC-220 — Specified dose on specified days
  Other Names: Iberdomide
Drug: Dexamethasone — Specified dose on specified days
  Other Names: Decadron
  Arms: Cohort B: CC-220 in combination with Dexamethasone (DEX) - Part 1; Cohort D: CC-220 in combination with Dexamethasone - Part 2; Cohort E: CC-220 with DEX and daratumumab (DARA) - Part 1; Cohort F: CC-220 with DEX and bortezomib - Part 1; Cohort G1: CC-220 in combination with CFZ and DEX - Part 1; Cohort G2 - CC-220 in combination with CFZ and DEX - Part 1; Cohort I: CC-220 in combination with DEX in post BCMA RRMM - Part 2; Cohort J1: CC-220 in combination with DEX and BTZ in NDMM - Part 2; Cohort J2: CC-220 in combination with DEX and BTZ in NDMM - Part 2; Cohort K: CC-220 with DEX and DARA in NDMM and not autologous stem cell transplant eligible - Part 2
Drug: Daratumumab — Specified dose on specified days
  Other Names: Darzalex
  Arms: Cohort E: CC-220 with DEX and daratumumab (DARA) - Part 1; Cohort K: CC-220 with DEX and DARA in NDMM and not autologous stem cell transplant eligible - Part 2
Drug: Bortezomib — Specified dose on specified days
  Other Names: Velcade
  Arms: Cohort F: CC-220 with DEX and bortezomib - Part 1; Cohort J1: CC-220 in combination with DEX and BTZ in NDMM - Part 2; Cohort J2: CC-220 in combination with DEX and BTZ in NDMM - Part 2
Drug: Carfilzomib — Specified dose on specified days
  Other Names: Kyprolis
  Arms: Cohort G1: CC-220 in combination with CFZ and DEX - Part 1; Cohort G2 - CC-220 in combination with CFZ and DEX - Part 1

SUMMARY:
This is a multicenter, multi-country, open-label, Phase 1b/2a dose-escalation study consisting of two parts: dose escalation (Part 1) for CC-220 monotherapy, CC-220 in combination with DEX, CC-220 in combination with DEX and DARA, CC-220 in combination with DEX and BTZ and CC-220 in combination with DEX and CFZ; and the expansion of the RP2D (Part 2) for CC-220 monotherapy and CC-220 in combination with DEX for Relapsed Refractory Multiple Myeloma (RRMM), CC-220 in combination with DEX and BTZ, and CC-220 in combination with DEX and DARA for Newly Diagnosed Multiple Myeloma (NDMM).

DETAILED DESCRIPTION:
Subjects assigned to CC-220 monotherapy, who develop progressive disease (PD) will have the option to receive DEX in addition to CC-220 after consultation with the Medical Monitor. The dose of CC-220 will not be higher than the dose of CC-220 used in combination with dexamethasone in Cohort B that has been determined to be safe. Progressive disease must be confirmed in accordance with international myeloma working group (IMWG) criteria.

For Cohorts A and B, the starting dose level of CC-220, dose level 1, is 0.3 mg. A dose level -1, of 0.15 mg, may also be evaluated if the starting dose level of 0.3 mg for 21 days of a 28-day cycle is not tolerated. For Cohorts E and F, the starting dose level of CC-220, dose level 1, is one dose level below the maximum dose for Cohort B that has been determined to be safe by the dose escalation committee (DEC) at the start of enrollment for both cohorts. For Cohort E in addition to CC-220 and DEX, daratumumab will be administered intravenously (IV) at a 16mg/kg dose. For Cohort F in addition to CC-220 and DEX, bortezomib will be administered subcutaneous (SC) at a 1.3mg/m2 dose.

All subjects who discontinue study treatment in Part 1 or Part 2 of the study for a reason other than PD or withdrawal of consent from the study will be followed for response assessment every 28 days (every 21 days for Cohort F) until PD.

The study will be conducted in compliance with the International Council for Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

The initiation of Part 2 will begin when the recommended phase 2 dose (RP2D) is established in Part 1 in either Cohort A, Cohort B, Cohort E or Cohort F. The cohorts may begin once the RP2D is determined for each cohort independently during Part 1. All expansion decisions will be determined by the DEC after review of all safety, PK, biomarker and preliminary efficacy data, as applicable. During Part 2, the Independent Expert Reviewer will review safety data and any other data deemed relevant so that subject safety is ensured.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2
* Relapsed and refractory multiple myeloma (RRMM) participants must have documented disease progression on or within 60 days from the last dose of their last myeloma therapy
* Newly diagnosed multiple myeloma (NDMM) participants must have documented diagnosis with previously untreated symptomatic multiple myeloma (MM)
* Participants in Cohorts J1 and K are those for whom autologous stem cell transplantation is not planned for initial therapy or are not considered by the investigator as eligible for high-dose chemotherapy and autologous stem cell transplantation

Exclusion Criteria:

* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study
* Nonsecretory multiple myeloma
* Prior history of malignancies, other than MM and select non-invasive malignancies, unless the participant has been free of the disease for ≥ 5 years

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2028-02-06 (Estimated)

PRIMARY OUTCOMES:
Establish maximum tolerated doses (MTDs) of CC-220 as monotherapy and in combination with other treatment | Approximately 3 years
  Establish the maximum tolerated doses (MTDs) of CC-220 monotherapy, in combination with DEX, and in combination with DEX and daratumumab (CC-220Dd), in combination with DEX and bortezomib (CC-220Vd), and in combination with DEX and carfilzomib (CC-220Kd)
Establish Recommended Phase 2 doses (RP2Ds) of CC-220 as monotherapy and in combination with other treatment | Approximately 3 years
  RP2D is defined as the dose selected for phase 2 based on safety, pharmacokinetics and biomarker data from phase 1 of the study
Overall response rate (ORR) of CC-220 in combination with Dexamethasone (DEX) in Cohort D | Approximately 5 years
  Tumor response, including progressive disease (PD) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria (Kumar, 2011) in CC-220 in combination with DEX

SECONDARY OUTCOMES:
Adverse Events (AEs) | Approximately 5 years
  Type, frequency, seriousness and severity of adverse events (AEs) (and AEs of special interest) and relationship of AEs to investigational product
Overall response rate (ORR) | Approximately 5 years
  Tumor response, including progressive disease (PD) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria (Kumar, 2016) for subjects who achieved partial response (PR) or better
Time to Response (TTR) | Approximately 5 years
  Is defined as the time from the first date of dosing of IP to the first date of documented response (partial response [PR] or greater)
Duration of Response (DOR) | Approximately 5 years
  Is defined as Time from the first documentation of response (PR or greater) to the first documentation of Progressive disease (PD)
Progression-free Survival (PFS) | Approximately 5 years
  Time from the first dose of investigational product (IP) to the first documentation of PD or death from any cause, whichever occurs first
Overall Survival (OS) in Part 2 relapsed and refractory multiple myeloma (RRMM) cohorts | Approximately 5 years
  Time from first dose of IP to death due to any cause
Pharmacokinetics - Area under the plasma concentration-time curve from time zero to tau, where tau is the dosing interval (AUC[TAU]) | Approximately 1 year
Pharmacokinetics - Maximum plasma concentration of drug (Cmax) | Approximately 1 year
Pharmacokinetics - Time to maximum plasma concentration of drug (Tmax) | Approximately 1 year
Very good partial response or better rate (VGPR) | Approximately 4 years
  Tumor response, including progressive disease (PD) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria (Kumar, 2016) for subjects who achieved VGPR or better

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (89):
- United States (34):
  - Local Institution - 102, Scottsdale, Arizona
  - Local Institution - 107, Little Rock, Arkansas
  - Local Institution - 101, Atlanta, Georgia
  - Local Institution - 120, Chicago, Illinois
  - Local Institution - 113, Fairway, Kansas
  - Local Institution - 106, Baltimore, Maryland
  - Local Institution - 114, Boston, Massachusetts
  - Local Institution - 115, Boston, Massachusetts
  - Local Institution - 110, Boston, Massachusetts
  - Local Institution - 104, Ann Arbor, Michigan
  - Local Institution - 103, Detroit, Michigan
  - Local Institution - 140, Grand Island, Nebraska
  - Local Institution - 141, Grand Island, Nebraska
  - Local Institution - 137, Omaha, Nebraska
  - Local Institution - 138, Omaha, Nebraska
  - Local Institution - 131, Omaha, Nebraska
  - Local Institution - 139, Papillion, Nebraska
  - Local Institution - 756, Cherry Hill, New Jersey
  - Local Institution - 108, Hackensack, New Jersey
  - Local Institution - 122, Mineola, New York
  - Local Institution - 121, New York, New York
  - Local Institution - 109, New York, New York
  - Local Institution - 111, New York, New York
  - Local Institution - 125, Rochester, New York
  - Local Institution - 112, Charlotte, North Carolina
  - Local Institution - 117, Cleveland, Ohio
  - Local Institution - 124, Columbus, Ohio
  - Local Institution - 116, Philadelphia, Pennsylvania
  - Local Institution - 123, Greenville, South Carolina
  - Local Institution - 134, Memphis, Tennessee
  - Local Institution - 118, Dallas, Texas
  - Local Institution - 119, Salt Lake City, Utah
  - Local Institution - 126, Seattle, Washington
  - Local Institution - 132, Tacoma, Washington
- Australia (2):
  - Local Institution - 854, Adelaide, South Australia
  - Local Institution - 852, Box Hill, Victoria
- Canada (4):
  - Local Institution - 904, Calgary, Alberta
  - Local Institution - 901, Vancouver, British Columbia
  - Local Institution - 902, Halifax, Nova Scotia
  - Local Institution - 903, Montreal, Quebec
- France (4):
  - Local Institution - 704, Lile Cedax
  - Local Institution - 701, Pessac
  - Local Institution - 703, Pierre-Bénite
  - Local Institution - 702, Poitiers
- Germany (6):
  - Local Institution - 605, Dresden
  - Local Institution - 603, Düsseldorf
  - Local Institution - 604, Hamburg
  - Local Institution - 602, Heidelberg
  - Local Institution - 601, Tübingen
  - Local Institution - 606, Würzburg
- Israel (3):
  - Local Institution - 751, Jerusalem, Jerusalem
  - Local Institution - 755, Tel Aviv
  - Local Institution - 754, Tel Litwinsky
- Italy (5):
  - Local Institution - 307, Meldola
  - Local Institution - 305, Pavia
  - Local Institution - 302, Reggio Emilia
  - Local Institution - 303, Rome
  - Local Institution - 301, Torino
- Japan (15):
  - Local Institution - 808, Matsuyama, Ehime
  - Local Institution - 805, Aomori
  - Local Institution - 813, Hiroshima
  - Local Institution - 812, Isehara City, Kanagawa
  - Local Institution - 809, Kamogawa
  - Local Institution - 802, Kyoto
  - Local Institution - 811, Nagasaki
  - Local Institution - 810, Nagoya
  - Local Institution - 801, Nagoya
  - Local Institution - 804, Osaka
  - Local Institution - 815, Ōgaki
  - Local Institution - 803, Sendai
  - Local Institution - 806, Shinagawa-ku, Tokyo
  - Local Institution - 814, Sunto-gun
  - Local Institution - 807, Toyohashi
- Netherlands (4):
  - Local Institution - 503, Amsterdam, North Holland
  - Local Institution - 504, Maastrich
  - Local Institution - 501, Rotterdam
  - Local Institution - 502, Utrecht
- Spain (7):
  - Local Institution - 404, Badalona (Barcelona)
  - Local Institution - 401, Barcelona
  - Local Institution - 405, Barcelona
  - Local Institution - 408, Madrid
  - Local Institution - 407, Madrid
  - Local Institution - 402, Pamplona
  - Local Institution - 406, Valencia
- United Kingdom (5):
  - Local Institution - 205, Birmingham
  - Local Institution - 202, Leeds
  - Local Institution - 204, Oxford
  - Local Institution - 201, Sutton
  - Local Institution - 203, Sutton

REFERENCES:
- [Derived] Amatangelo M, Flynt E, Stong N, Ray P, Van Oekelen O, Wang M, Ortiz M, Maciag P, Peluso T, Parekh S, van de Donk NWCJ, Lonial S, Thakurta A. Pharmacodynamic changes in tumor and immune cells drive iberdomide's clinical mechanisms of activity in relapsed and refractory multiple myeloma. Cell Rep Med. 2024 Jun 18;5(6):101571. doi: 10.1016/j.xcrm.2024.101571. Epub 2024 May 21. PMID 38776914
- [Derived] Lonial S, Popat R, Hulin C, Jagannath S, Oriol A, Richardson PG, Facon T, Weisel K, Larsen JT, Minnema MC, Abdallah AO, Badros AZ, Knop S, Stadtmauer EA, Cheng Y, Amatangelo M, Chen M, Nguyen TV, Amin A, Peluso T, van de Donk NWCJ. Iberdomide plus dexamethasone in heavily pretreated late-line relapsed or refractory multiple myeloma (CC-220-MM-001): a multicentre, multicohort, open-label, phase 1/2 trial. Lancet Haematol. 2022 Nov;9(11):e822-e832. doi: 10.1016/S2352-3026(22)00290-3. Epub 2022 Oct 6. PMID 36209764
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT02773030.html